CLINICAL TRIAL: NCT03955471
Title: A Phase 2 Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of the Combination of Niraparib and Dostarlimab (TSR-042) in Patients With Platinum-Resistant Ovarian Cancer (MOONSTONE)
Brief Title: Study to Evaluate the Efficacy and Safety of the Combination of Niraparib and Dostarlimab (TSR-042) in Participants With Platinum Resistant Ovarian Cancer
Acronym: MOONSTONE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study will not resume based on the results of a planned interim analysis that showed futility
Sponsor: Tesaro, Inc. (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213353; 3000-02-006 (Other: Tesaro)
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Neoplasms
Keywords: Open-label; Single-arm; Efficacy and Safety; Platinum-resistant ovarian cancer; Niraparib; dostarlimab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib+Dostarlimab (TSR-042) (Experimental): Participants with body weight ≥77 kilogram (kg) and platelet count ≥150,000/microliter (μL) at baseline were administered Niraparib 300 milligram (mg) once daily (QD) and participants with body weight <77 kg or platelet count <150,000/μL at baseline were administered Niraparib 200 mg QD. Niraparib was administered continuously until Progressive disease (PD) or toxicity. Dostarlimab (TSR-042) was administered as an intravenous (IV) infusion of 500 mg once every three weeks (Q3W) from Cycle 1 Day 1 through Cycle 4. Beginning at Cycle 5, Dostarlimab (TSR-042) was administered via an IV infusion of 1000 mg on Day 1 of each 6-week cycle until PD or toxicity, up to 27 months.
  Interventions: Drug: Niraparib; Drug: Dostarlimab

INTERVENTIONS:
Drug: Niraparib — Niraparib is a potent, orally active poly (adenosine diphosphate-ribose) polymerase (PARP)-1 and PARP2 inhibitor being developed as a treatment for participants with tumors that harbor defects in the homologous recombination deoxyribonucleic acid (DNA) repair pathway or that are driven by PARP-mediated transcription factors.
  Other Names: ZEJULA
Drug: Dostarlimab — TSR-042 is a humanized monoclonal antibody that binds with high affinity to programmed cell death-1 (PD-1) resulting in inhibition of binding to programmed cell-death receptor ligands 1 and 2 (PD-L1 and PD-L2).

SUMMARY:
This is an open-label, single-arm Phase 2 study to evaluate the efficacy and safety of combination of niraparib and dostarlimab (TSR-042) in participants with advanced, relapsed, high-grade ovarian, fallopian tube, endometrioid, clear cell ovarian or primary peritoneal cancer without known breast cancer susceptibility gene (BRCA) mutation who have platinum-resistant disease and who have also been previously treated with bevacizumab.

ELIGIBILITY:
Inclusion criteria:

* Participant must be female >=18 years of age, able to understand the study procedures, and subsequently agreed to participate in the study by providing written informed consent.
* Participants must have recurrent high-grade serous, endometrioid, or clear cell ovarian, fallopian tube, or primary peritoneal cancer.
* Participants must be considered resistant to the last administered platinum therapy.
* Participants must have completed at least 1 but no more than 3 prior lines of therapy for advanced or metastatic ovarian cancer.
* Participants must have been previously treated with platinum-based regimen, taxane agent(s), and bevacizumab.
* Participant has measurable disease according to RECIST v.1.1.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant has adequate organ function.
* Females with childbearing potential have a serum pregnancy test that is negative 72 prior first dose and are not breastfeeding. Participant must also agree to abstain from activities that could result in pregnancy from enrollment through 180 days after the last dose of study treatment.
* Participant must provide formalin fixed paraffin embedded (FFPE) tumor tissue block(s) with sufficient tumor content (as confirmed by the Sponsor's designated central laboratory) during screening to enable BRCA testing and PD-L1 testing. The use of slides created from paraffin-embedded tissue as opposed to FFPE blocks must be approved by the Sponsor.
* Participant must agree to complete health-related quality of life (HRQoL) questionnaires throughout the study.

Exclusion Criteria:

* Participant who experienced disease progression within 3 months (12 weeks or 84 days) of first-line platinum therapy.
* Participants with a known deleterious or suspected BRCA 1 or 2 mutation.
* Participant has received prior therapy with an anti-PD-1, anti-PD-L1 or anti-PD-L2 agent.
* Participant has received prior therapy with a PARP-1/PARP-2 inhibitor.
* Participant has a known hypersensitivity to dostarlimab (TSR-042), Niraparib, their components, or their excipients.
* Participant has a known history of myelodysplastic syndrome or acute myeloid leukemia.
* Participant has not recovered from prior chemotherapy induced adverse events.
* Participant has a known diagnosis of immunodeficiency or is receiving systemic steroid therapy exceeding an equivalent of prednisone 10 mg daily or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Participant is currently participating in a treatment study or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment.
* Participant has received prior systemic anticancer therapy including cytotoxic chemotherapy, hormonal therapy given with the intention to treat ovarian cancer, or biological therapy within 3 weeks of the first dose of study treatment.
* Participant has received live vaccine within 14 days of planned start of study therapy
* Participant has symptomatic uncontrolled brain or leptomeningeal metastases. (If investigator feels participant symptoms are not symptomatic, participants can undergo a scan to confirm for eligibility).
* Participant had major surgery with 4 weeks of starting the first dose of the study treatment or participant has not recovered from any effects of any major surgery.
* Participant has a known additional malignancy that progressed or required active treatment within the last 2 years.
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active controlled infection.
* Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study.
* Participant has known active hepatitis B (hepatitis B surface antigen reactive) or hepatitis C (hepatitis C virus ribonucleic acid, qualitative).
* Participant with a known history of human immunodeficiency virus (HIV) are allowed if they meet all of the following criteria:

  1. Cluster of differentiation 4 >=350/microliter (μL) and viral load <400 copies/milliliter (mL)
  2. No history of acquired immunodeficiency syndrome-defining opportunistic infections within 12 months prior to enrollment
  3. No history of HIV-associated malignancy for the past 5 years
  4. Concurrent antiretroviral therapy as per the most current National Institutes of Health (NIH) Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV started >4 weeks prior to study enrollment
* Participant is immunocompromised. Participants with splenectomy are allowed.
* Participant has an ongoing bowel obstruction or has other conditions that would lead to impaired absorption of oral niraparib.
* Participant has active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (25):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Solvang, California
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Randall LM, O'Malley DM, Monk BJ, Coleman RL, Gaillard S, Adams S, Duska LR, Dalton H, Holloway RW, Huang M, Chon HS, Cloven NG, ElNaggar AC, O'Cearbhaill RE, Waggoner S, Tarkar A, Striha A, Nelsen LM, Baines A, Samnotra V, Konstantinopoulos PA. Niraparib and dostarlimab for the treatment of recurrent platinum-resistant ovarian cancer: results of a Phase II study (MOONSTONE/GOG-3032). Gynecol Oncol. 2023 Nov;178:161-169. doi: 10.1016/j.ygyno.2023.10.005. Epub 2023 Oct 25. PMID 37890345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2019 until September 2020, 72 participants were screened and 41 participants were enrolled (31 screen failures)
Pre-assignment Details: This study was terminated as the interim analysis of the primary endpoint met the prespecified futility criteria.
Period: Overall Study
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Started | 41
Completed | 1
Not Completed | 40
Not completed — Death | 22
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6
Not completed — Sponsor Decision to Terminate Study | 11

BASELINE CHARACTERISTICS:
Groups:
- Niraparib+Dostarlimab (TSR-042): Participants with body weight ≥77 kg and platelet count ≥150,000/μL at baseline were administered Niraparib 300 mg QD and participants with body weight <77 kg or platelet count <150,000/μL at baseline were administered Niraparib 200 mg QD. Niraparib was administered continuously until PD or toxicity. Dostarlimab (TSR-042) was administered as an IV infusion of 500 mg Q3W from Cycle 1 Day 1 through Cycle 4. Beginning at Cycle 5, Dostarlimab was administered via an IV infusion of 1000 mg on Day 1 of each 6-week cycle until PD or toxicity, up to 27 months.
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 62.9 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Black or African American | 3
  Unknown | 3
  White | 32

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Participants With Platinum-resistant Ovarian Cancer (PROC)
Description: ORR is defined as the percentage of participants who have achieved confirmed complete response (CR) or partial response (PR), as determined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) criteria based on Investigator assessment and computed tomography (CT) scans were commonly used for tumor imaging.
Time Frame: Up to approximately 22 months
Population: Safety (SAF) Population: All participants who receive any amount of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Percentage of Participants | 7.3 [1.5 to 19.9]

2. Primary Outcome: ORR in Participants With PROC Who Have Programmed Cell Death-ligand 1 (PD-L 1) Positive Status
Description: ORR is defined as the percentage of participants who have achieved confirmed CR or PR, as determined by RECIST v1.1 criteria based on Investigator assessment and CT scans were commonly used for tumor imaging. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with combined positive score (vCPS) >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data for participants with PD-L1 positive status in the SAF population are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 13
Percentage of Participants | 7.7 [0.2 to 36]

3. Secondary Outcome: Duration of Response (DOR) in Participants With PROC
Description: DOR is defined as the time from first documentation of response (CR or PR) until the time of first documentation of disease progression or death by any cause in the absence of progression by RECIST v.1.1 based on Investigator assessment.
Time Frame: Up to approximately 22 months
Population: SAF Population. DOR has been summarized only for responders.
Measure: Median (Full Range); unit: Months
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 3
Months | 3.8 [3 to 9.2]

4. Secondary Outcome: DOR in Participants With PROC Who Have PD-L 1 Positive Status
Description: DOR is defined as the time from first documentation of response (CR or PR) until the time of first documentation of disease progression or death by any cause in the absence of progression by RECIST v.1.1 based on Investigator assessment. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with vCPS >=5% was used as specified cut-point for the assessment of PD-L1 patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data for participants with PD-L1 positive status in the SAF population are presented. DOR has been summarized only for responders.
Measure: Median (Full Range); unit: Months
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 1
Months | NA [3.8 to NA] — The Median and Upper Limit was not estimable due to low number of participants with PD-L1 positive status.

5. Secondary Outcome: Progression-free Survival (PFS) in Participants With PROC
Description: PFS is defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression by RECIST v.1.1 based on Investigator assessment.
Time Frame: Up to approximately 22 months
Population: SAF Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Months | 2.1 [1.97 to 2.23]

6. Secondary Outcome: PFS in Participants With PROC Who Have PD-L 1 Positive Status
Description: PFS is defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression by RECIST v.1.1 based on Investigator assessment. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with a vCPS >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data for participants with PD-L1 positive status in the SAF population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 13
Months | 2.22 [1.64 to NA] — The upper limit of the 95% CI was not estimable due to limited number of events.

7. Secondary Outcome: Overall Survival (OS) in Participants With PROC
Description: OS is defined as the time from the date of the first dose of study treatment to the date of death by any cause.
Time Frame: Up to approximately 22 months
Population: SAF Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Months | 10.61 [7.26 to 13.44]

8. Secondary Outcome: OS in Participants With PROC Who Have PD-L 1 Positive Status
Description: OS is defined as the time from the date of the first dose of study treatment to the date of death by any cause. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with vCPS >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data for participants with PD-L1 positive status in the SAF population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 13
Months | NA [7.26 to NA] — The median and upper limit of the 95% CI was not estimable due to limited number of events.

9. Secondary Outcome: Disease Control Rate (DCR) in Participants With PROC
Description: DCR is defined as the percentage of participants who have achieved best overall response (BOR) of CR, PR, or stable disease (SD) per RECIST v.1.1 based on the investigator's assessment.
Time Frame: Up to approximately 22 months
Population: SAF Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Percentage of Participants | 29.3 [16.1 to 45.5]

10. Secondary Outcome: DCR in Participants With PROC Who Have PD-L 1 Positive Status
Description: DCR is defined as the percentage of participants who have achieved BOR of CR, PR, or SD per RECIST v.1.1 based on the investigator's assessment. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with vCPS >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data for participants with PD-L1 positive status in the SAF population are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 13
Percentage of Participants | 38.5 [13.9 to 68.4]

11. Secondary Outcome: ORR in Participants With PROC Based on Independent Review Committee (IRC) Assessment
Description: ORR is defined as the percentage of participants who have achieved confirmed CR or PR per RECIST v1.1 based on the independent review committee assessment.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination.
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

12. Secondary Outcome: ORR in Participants With PROC Who Have PD-L 1 Positive Status Based on IRC Assessment
Description: ORR is defined as the percentage of participants who have achieved confirmed CR or PR per RECIST v1.1 based on the independent review committee assessment. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with a vCPS >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

13. Secondary Outcome: DOR in Participants With PROC Based on IRC Assessment
Description: DOR is defined as the time from first documentation of response (CR or PR) until the time of first documentation of disease progression or death by any cause in the absence of progression by RECIST v.1.1 based on Independent Review Committee assessment.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

14. Secondary Outcome: DOR in Participants With PROC Who Have PD-L 1 Positive Status Based on IRC Assessment
Description: DOR is defined as the time from first documentation of response (CR or PR) until the time of first documentation of disease progression or death by any cause in the absence of progression by RECIST v.1.1 based on Independent Review Committee assessment. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with a vCPS >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

15. Secondary Outcome: PFS in Participants With PROC Based on IRC Assessment
Description: PFS is defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression by RECIST v.1.1 based on Independent Review Committee Assessment.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

16. Secondary Outcome: PFS in Participants With PROC Who Have PD-L 1 Positive Status Based on IRC Assessment
Description: PFS is defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression by RECIST v.1.1 based on IRC Assessment. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with a vCPS >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

17. Secondary Outcome: DCR in Participants With PROC Based on IRC Assessment
Description: DCR is defined as the percentage of participants who have achieved BOR of CR, PR, or SD per RECIST v.1.1 based on IRC Assessment.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

18. Secondary Outcome: DCR in Participants With PROC Who Have PD-L 1 Positive Status Based on IRC Assessment
Description: DCR is defined as the percentage of participants who have achieved BOR of CR, PR, or SD per RECIST v.1.1 based on Independent Review Committee Assessment. PD-L1 is a ligand that binds to PD-L1 protein on tumor infiltrating T cells and renders the T cells inactive. Any PD-L1 positive tissue sample with vCPS >=5% was used as specified cut-point for the assessment of PD-L1 positive patient subset with PROC. vCPS was defined as the percentage of tumor cells and immune cells staining positive within the total tumor area.
Time Frame: Up to approximately 22 months
Population: Data was not collected as IRC assessment was not utilized due to study termination
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 0

19. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-emergent Adverse Events (TEAEs) and Adverse Event of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a patient administered with a medicinal product and that does which may or may not have a causal relationship with this treatment. A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. TEAEs are any event that occurred between first dose of study drug up to 22 months, which were absent before treatment or that had worsened relative to pretreatment state. AESI were any AE (serious or non-serious) that is of scientific and medical concern specific to the study treatment, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was done.
Time Frame: Up to approximately 27 months
Population: SAF Population
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Participants
  AEs | 41
  SAEs | 23
  TEAE | 41
  AESIs | 2

20. Secondary Outcome: Number of Participants With Grade Shift From Baseline in Hematology
Description: Blood samples were collected for the analysis of hematology parameters and each parameter was graded according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.3. Grade 0: Normal, Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent measurement prior to the first administration of study treatment. Data has been presented for the number of participants with hematology grade shifts from baseline grade to grade 3 and 4 for each parameter.
Time Frame: Up to approximately 27 months
Population: SAF Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Participants
  Hemoglobin, Grade 0 to Grade 3 | 3
  Hemoglobin, Grade 1 to Grade 3 | 5
  Hemoglobin, Grade 2 to Grade 3 | 1
  Hemoglobin, Grade 3 to Grade 3 | 0
  Hemoglobin, Grade 4 to Grade 3 | 0
  Hemoglobin, Grade 0 to Grade 4 | 0
  Hemoglobin, Grade 1 to Grade 4 | 0
  Hemoglobin, Grade 2 to Grade 4 | 0
  Hemoglobin, Grade 3 to Grade 4 | 0
  Hemoglobin, Grade 4 to Grade 4 | 0
  Leukocytes, Grade 0 to Grade 3 | 0
  Leukocytes, Grade 1 to Grade 3 | 0
  Leukocytes, Grade 2 to Grade 3 | 0
  Leukocytes, Grade 3 to Grade 3 | 0
  Leukocytes, Grade 4 to Grade 3 | 0
  Leukocytes, Grade 0 to Grade 4 | 0
  Leukocytes, Grade 1 to Grade 4 | 0
  Leukocytes, Grade 2 to Grade 4 | 0
  Leukocytes, Grade 3 to Grade 4 | 0
  Leukocytes, Grade 4 to Grade 4 | 0
  Lymphocytes, Grade 0 to Grade 3 | 5
  Lymphocytes, Grade 1 to Grade 3 | 3
  Lymphocytes, Grade 2 to Grade 3 | 3
  Lymphocytes, Grade 3 to Grade 3 | 0
  Lymphocytes, Grade 4 to Grade 3 | 0
  Lymphocytes, Grade 0 to Grade 4 | 1
  Lymphocytes, Grade 1 to Grade 4 | 0
  Lymphocytes, Grade 2 to Grade 4 | 0
  Lymphocytes, Grade 3 to Grade 4 | 0
  Lymphocytes, Grade 4 to Grade 4 | 0
  Neutrophil Count, Grade 0 to Grade 3 | 1
  Neutrophil Count, Grade 1 to Grade 3 | 0
  Neutrophil Count, Grade 2 to Grade 3 | 0
  Neutrophil Count, Grade 3 to Grade 3 | 0
  Neutrophil Count, Grade 4 to Grade 3 | 0
  Neutrophil Count, Grade 0 to Grade 4 | 1
  Neutrophil Count, Grade 1 to Grade 4 | 0
  Neutrophil Count, Grade 2 to Grade 4 | 0
  Neutrophil Count, Grade 3 to Grade 4 | 0
  Neutrophil Count, Grade 4 to Grade 4 | 0
  Platelets, Grade 0 to Grade 3 | 4
  Platelets, Grade 1 to Grade 3 | 1
  Platelets, Grade 2 to Grade 3 | 0
  Platelets, Grade 3 to Grade 3 | 0
  Platelets, Grade 4 to Grade 3 | 0
  Platelets, Grade 0 to Grade 4 | 4
  Platelets, Grade 1 to Grade 4 | 0
  Platelets, Grade 2 to Grade 4 | 0
  Platelets, Grade 3 to Grade 4 | 0
  Platelets, Grade 4 to Grade 4 | 0

21. Secondary Outcome: Number of Participants With Grade Shift From Baseline in Plasma Chemistry
Description: Blood samples were collected and the clinical chemistry parameters assessed were Albumin (Alb), alanine aminotransferase (ALT), amylase, aspartate aminotransferase (AST), alkaline phosphatase (ALP), sodium, total bilirubin (TB), creatinine, glucose, magnesium and potassium. The Grade shift post baseline data of each parameter from Grade 0 through Grade 4 was based on the CTCAE version 4.03, grading scale, as per intensity, namely Grade 0: Normal, Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent measurement prior to the first administration of study treatment. Data has been presented for the number of participants with plasma chemistry grade shifts from baseline grade to grade 3 and 4 for each parameter.
Time Frame: Up to approximately 27 months
Population: SAF Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Participants
  ALT, Grade 0 to Grade 3 | 3
  ALT, Grade 1 to Grade 3 | 0
  ALT, Grade 2 to Grade 3 | 0
  ALT, Grade 3 to Grade 3 | 0
  ALT, Grade 4 to Grade 3 | 0
  ALT, Grade 0 to Grade 4 | 1
  ALT, Grade 1 to Grade 4 | 0
  ALT, Grade 2 to Grade 4 | 0
  ALT, Grade 3 to Grade 4 | 0
  ALT, Grade 4 to Grade 4 | 0
  Alb, Grade 0 to Grade 3 | 1
  Alb, Grade 1 to Grade 3 | 0
  Alb, Grade 2 to Grade 3 | 0
  Alb, Grade 3 to Grade 3 | 0
  Alb, Grade 4 to Grade 3 | 0
  Alb, Grade 0 to Grade 4 | 0
  Alb, Grade 1 to Grade 4 | 0
  Alb, Grade 2 to Grade 4 | 0
  Alb, Grade 3 to Grade 4 | 0
  Alb, Grade 4 to Grade 4 | 0
  ALP, Grade 0 to Grade 3 | 3
  ALP, Grade 1 to Grade 3 | 1
  ALP, Grade 2 to Grade 3 | 1
  ALP, Grade 3 to Grade 3 | 0
  ALP, Grade 4 to Grade 3 | 0
  ALP, Grade 0 to Grade 4 | 0
  ALP, Grade 1 to Grade 4 | 1
  ALP, Grade 2 to Grade 4 | 0
  ALP, Grade 3 to Grade 4 | 0
  ALP, Grade 4 to Grade 4 | 0
  Amylase, Grade 0 to Grade 3 | 0
  Amylase, Grade 1 to Grade 3 | 0
  Amylase, Grade 2 to Grade 3 | 0
  Amylase, Grade 3 to Grade 3 | 0
  Amylase, Grade 4 to Grade 3 | 0
  Amylase, Grade 0 to Grade 4 | 0
  Amylase, Grade 1 to Grade 4 | 0
  Amylase, Grade 2 to Grade 4 | 0
  Amylase, Grade 3 to Grade 4 | 0
  Amylase, Grade 4 to Grade 4 | 0
  AST, Grade 0 to Grade 3 | 4
  AST, Grade 1 to Grade 3 | 1
  AST, Grade 2 to Grade 3 | 0
  AST, Grade 3 to Grade 3 | 0
  AST, Grade 4 to Grade 3 | 0
  AST, Grade 0 to Grade 4 | 0
  AST, Grade 1 to Grade 4 | 0
  AST, Grade 2 to Grade 4 | 0
  AST, Grade 3 to Grade 4 | 0
  AST, Grade 4 to Grade 4 | 0
  TB, Grade 0 to Grade 3 | 1
  TB, Grade 1 to Grade 3 | 0
  TB, Grade 2 to Grade 3 | 0
  TB, Grade 3 to Grade 3 | 0
  TB, Grade 4 to Grade 3 | 0
  TB, Grade 0 to Grade 4 | 1
  TB, Grade 1 to Grade 4 | 0
  TB, Grade 2 to Grade 4 | 0
  TB, Grade 3 to Grade 4 | 0
  TB, Grade 4 to Grade 4 | 0
  Creatinine, Grade 0 to Grade 3 | 1
  Creatinine, Grade 1 to Grade 3 | 0
  Creatinine, Grade 2 to Grade 3 | 0
  Creatinine, Grade 3 to Grade 3 | 0
  Creatinine, Grade 4 to Grade 3 | 0
  Creatinine, Grade 0 to Grade 4 | 0
  Creatinine, Grade 1 to Grade 4 | 0
  Creatinine, Grade 2 to Grade 4 | 0
  Creatinine, Grade 3 to Grade 4 | 0
  Creatinine, Grade 4 to Grade 4 | 0
  Glucose high, Grade 0 to Grade 3 | 0
  Glucose high, Grade 1 to Grade 3 | 3
  Glucose high, Grade 2 to Grade 3 | 0
  Glucose high, Grade 3 to Grade 3 | 1
  Glucose high, Grade 4 to Grade 3 | 0
  Glucose high, Grade 0 to Grade 4 | 0
  Glucose high, Grade 1 to Grade 4 | 0
  Glucose high, Grade 2 to Grade 4 | 0
  Glucose high, Grade 3 to Grade 4 | 0
  Glucose high, Grade 4 to Grade 4 | 0
  Glucose low, Grade 0 to Grade 3 | 0
  Glucose low, Grade 1 to Grade 3 | 0
  Glucose low, Grade 2 to Grade 3 | 0
  Glucose low, Grade 3 to Grade 3 | 0
  Glucose low, Grade 4 to Grade 3 | 0
  Glucose low, Grade 0 to Grade 4 | 0
  Glucose low, Grade 1 to Grade 4 | 0
  Glucose low, Grade 2 to Grade 4 | 0
  Glucose low, Grade 3 to Grade 4 | 0
  Glucose low, Grade 4 to Grade 4 | 0
  Magnesium high, Grade 0 to Grade 3 | 1
  Magnesium high, Grade 1 to Grade 3 | 0
  Magnesium high, Grade 2 to Grade 3 | 0
  Magnesium high, Grade 3 to Grade 3 | 0
  Magnesium high, Grade 4 to Grade 3 | 0
  Magnesium high, Grade 0 to Grade 4 | 0
  Magnesium high, Grade 1 to Grade 4 | 0
  Magnesium high, Grade 2 to Grade 4 | 0
  Magnesium high, Grade 3 to Grade 4 | 0
  Magnesium high, Grade 4 to Grade 4 | 0
  Magnesium low, Grade 0 to Grade 3 | 0
  Magnesium low, Grade 1 to Grade 3 | 0
  Magnesium low, Grade 2 to Grade 3 | 0
  Magnesium low, Grade 3 to Grade 3 | 1
  Magnesium low, Grade 4 to Grade 3 | 0
  Magnesium low, Grade 0 to Grade 4 | 0
  Magnesium low, Grade 1 to Grade 4 | 0
  Magnesium low, Grade 2 to Grade 4 | 0
  Magnesium low, Grade 3 to Grade 4 | 0
  Magnesium low, Grade 4 to Grade 4 | 0
  Potassium high, Grade 0 to Grade 3 | 0
  Potassium high, Grade 1 to Grade 3 | 0
  Potassium high, Grade 2 to Grade 3 | 0
  Potassium high, Grade 3 to Grade 3 | 0
  Potassium high, Grade 4 to Grade 3 | 0
  Potassium high, Grade 0 to Grade 4 | 0
  Potassium high, Grade 1 to Grade 4 | 0
  Potassium high, Grade 2 to Grade 4 | 0
  Potassium high, Grade 3 to Grade 4 | 0
  Potassium high, Grade 4 to Grade 4 | 0
  Potassium low, Grade 0 to Grade 3 | 3
  Potassium low, Grade 1 to Grade 3 | 1
  Potassium low, Grade 2 to Grade 3 | 0
  Potassium low, Grade 3 to Grade 3 | 0
  Potassium low, Grade 4 to Grade 3 | 0
  Potassium low, Grade 0 to Grade 4 | 0
  Potassium low, Grade 1 to Grade 4 | 0
  Potassium low, Grade 2 to Grade 4 | 0
  Potassium low, Grade 3 to Grade 4 | 0
  Potassium low, Grade 4 to Grade 4 | 0
  Sodium high, Grade 0 to Grade 3 | 0
  Sodium high, Grade 1 to Grade 3 | 0
  Sodium high, Grade 2 to Grade 3 | 0
  Sodium high, Grade 3 to Grade 3 | 0
  Sodium high, Grade 4 to Grade 3 | 0
  Sodium high, Grade 0 to Grade 4 | 0
  Sodium high, Grade 1 to Grade 4 | 0
  Sodium high, Grade 2 to Grade 4 | 0
  Sodium high, Grade 3 to Grade 4 | 0
  Sodium high, Grade 4 to Grade 4 | 0
  Sodium low, Grade 0 to Grade 3 | 4
  Sodium low, Grade 1 to Grade 3 | 7
  Sodium low, Grade 2 to Grade 3 | 0
  Sodium low, Grade 3 to Grade 3 | 0
  Sodium low, Grade 4 to Grade 3 | 0
  Sodium low, Grade 0 to Grade 4 | 0
  Sodium low, Grade 1 to Grade 4 | 0
  Sodium low, Grade 2 to Grade 4 | 0
  Sodium low, Grade 3 to Grade 4 | 0
  Sodium low, Grade 4 to Grade 4 | 0

22. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Baseline was defined as the most recent measurement prior to the first administration of study treatment. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. The minimum (min) and maximum (max) change from baseline values have been reported.
Time Frame: Up to approximately 27 months
Population: SAF Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Millimeters of mercury
  DBP, max change post baseline | 10.6 (10.07)
  DBP, min change post baseline | -5.8 (11.87)
  SBP, max change post baseline | 16.5 (23.01)
  SBP, min change post baseline | -12.5 (24.61)

23. Secondary Outcome: Change From Baseline in Pulse Rate
Description: as for outcome 22
Time Frame: Up to approximately 27 months
Population: SAF Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Beats per minute
  max change post baseline | 20.5 (14.71)
  min change post baseline | 1 (13.77)

24. Secondary Outcome: Change From Baseline in Temperature
Description: as for outcome 22
Time Frame: Up to approximately 27 months
Population: SAF Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 41
Degrees Celsius
  max change post baseline | 0.31 (0.421)
  min change post baseline | -0.35 (0.422)

25. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio
Description: Blood samples were collected to evaluate Prothrombin International Normalized Ratio (INR). Baseline was defined as the most recent measurement prior to the first administration of study treatment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to approximately 27 months
Population: SAF Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 2
Ratio
  Day 2: number analyzed (Participants) | 1
  Day 2 | 0.2
  Day 41: number analyzed (Participants) | 1
  Day 41 | 0.3
  Day 52: number analyzed (Participants) | 1
  Day 52 | 0.7

26. Secondary Outcome: Change in Baseline in Activated Partial Thromboplastin Time
Description: Blood samples were planned to be collected to evaluate activated partial thromboplastin time (APTT). Baseline was defined as the most recent measurement prior to the first administration of study treatment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to approximately 27 months
Population: SAF Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 1
Second
  Day 2 | 1
  Day 41 | 16.9

27. Secondary Outcome: Change From Baseline in Thyrotropin
Description: Blood samples were collected to evaluate thyrotropin at indicated time points. Baseline was defined as the most recent measurement prior to the first administration of study treatment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to approximately 27 months
Population: SAF Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliunits per liter (mU/L)
Arm/Group | Niraparib+Dostarlimab (TSR-042)
Number analyzed (Participants) | 15
Milliunits per liter (mU/L)
  Cycle 5 Day 1 | 8.074 (19.737)
  Cycle 7 Day 1: number analyzed (Participants) | 4
  Cycle 7 Day 1 | 12.79 (23.240)
  Cycle 9 Day 1: number analyzed (Participants) | 1
  Cycle 9 Day 1 | 2.596
  Cycle 11 Day 1: number analyzed (Participants) | 1
  Cycle 11 Day 1 | 2.517

ADVERSE EVENTS:
Time Frame: All cause mortality, non-SAEs and SAEs were collected from Day 1 up to approximately 27 months.
Arm/Group | Niraparib+Dostarlimab (TSR-042)
All-Cause Mortality (participants affected / at risk) | 22/41
Serious Adverse Events (participants affected / at risk) | 23/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib+Dostarlimab (TSR-042) (N=41)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib+Dostarlimab (TSR-042) (N=41)
Anaemia (Blood and lymphatic system disorders) | 18 (63)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (11)
Palpitations (Cardiac disorders) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 24 (35)
Vomiting (Gastrointestinal disorders) | 19 (28)
Abdominal pain (Gastrointestinal disorders) | 15 (24)
Constipation (Gastrointestinal disorders) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 11 (14)
Abdominal distension (Gastrointestinal disorders) | 9 (11)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Ascites (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 18 (25)
Oedema peripheral (General disorders) | 7 (8)
Pyrexia (General disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Blood creatinine increased (Investigations) | 10 (21)
Platelet count decreased (Investigations) | 11 (18)
Blood alkaline phosphatase increased (Investigations) | 10 (17)
Aspartate aminotransferase increased (Investigations) | 8 (14)
Alanine aminotransferase increased (Investigations) | 6 (12)
Neutrophil count decreased (Investigations) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (15)
Decreased appetite (Metabolism and nutrition disorders) | 9 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 6 (7)
Anxiety (Psychiatric disorders) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (12)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Hypertension (Vascular disorders) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT03955471/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03955471/SAP_001.pdf